CLINICAL TRIAL: NCT02404545
Title: A Randomized Study of the Utility of Composite Mesh Placement to Prevent Parastomal Hernia in Patients Undergoing Urinary Diversion With Ileal Conduit
Brief Title: Prevention of Parastomal Hernia by Mesh Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor stopped producing device
Sponsor: University of Miami (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20140277
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Parastomal Hernia
Keywords: Hernia; Mesh; Ileal conduit
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Ideal Conduit No Mesh (No Intervention): No mesh will be placed at the time of radical cystectomy and ileal conduit.
- Group 2 - Ileal Conduit with Mesh (Active Comparator): Ethicon Physiomesh will be placed at the time of radical cystectomy and ileal conduit.
  Interventions: Device: Ethicon Physiomesh

INTERVENTIONS:
Device: Ethicon Physiomesh — Ethicon Physiomesh will be paced at the time of radical cystectomy and ileal conduit.
  Arms: Group 2 - Ileal Conduit with Mesh

SUMMARY:
Concurrent placement of a mesh during formation of ileal conduit will decrease the incidence of parastomal hernia and associated complications.

DETAILED DESCRIPTION:
Subject to inclusion and exclusion criteria, patients will be randomized 1:1 to the control and intervention groups:

Randomization groups:

* Group 1 (control): Ileal Conduit
* Group 2 (intervention): Ileal conduit with concurrent mesh placement.

Ethicon PHYSIOMESH composite mesh will be utilized for this study. This is a composite mesh with a reduced polypropylene content. It is a widely used, commercially available hernia mesh, and its use and placement are simple and well described. The mesh will be placed at the time of radical cystectomy and ileal conduit. A small circle of mesh, the diameter of the ileal conduit, will be excised to allow for fitment around the ileal conduit. The mesh will be placed so that it encompasses the ileal conduit in a non-constricting manner, and will be sutured to the anterior abdominal wall. Product will be stored in a secure, sterile manner at the UMH operating room sterile supply room, and in accordance with institutional policies.

Patients from both groups will be followed up in a standard fashion. Follow up visits and clinical assessment will be at 6 weeks after surgery, 3 monthly during the first year, then every 6 months for at least 5 years. During each visit, patients will be clinically evaluated for the presence or absence of parastomal hernia, and any routine surveillance radiology imaging will be reviewed.

Parastomal hernia is clinically defined as an incisional hernia at the site of the ileal conduit stoma. This may be clinically apparent by examining the patient during performance of abdominal straining or Valsalva maneuver, or may be evident on radiology imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients eligible to undergo urinary diversion with ileal conduit.
2. Patients with the ability to understand and willingness to sign a written informed consent document.
3. Men and Women aged 18 to 80 years.

Exclusion Criteria:

1. Patients unable or unwilling to consent to the proposed surgery
2. Pregnant women
3. Patients with prior ileal conduit surgery undergoing revision.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murugesan Manoharan, MD, Principal Investigator — University of Miami
Locations (1):
- University Of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carne PW, Robertson GM, Frizelle FA. Parastomal hernia. Br J Surg. 2003 Jul;90(7):784-93. doi: 10.1002/bjs.4220. PMID 12854101
- [Result] Israelsson LA. Preventing and treating parastomal hernia. World J Surg. 2005 Aug;29(8):1086-9. doi: 10.1007/s00268-005-7973-z. PMID 15981038
- [Result] Kouba E, Sands M, Lentz A, Wallen E, Pruthi RS. Incidence and risk factors of stomal complications in patients undergoing cystectomy with ileal conduit urinary diversion for bladder cancer. J Urol. 2007 Sep;178(3 Pt 1):950-4. doi: 10.1016/j.juro.2007.05.028. Epub 2007 Jul 16. PMID 17632147
- [Result] Pearl RK. Parastomal hernias. World J Surg. 1989 Sep-Oct;13(5):569-72. doi: 10.1007/BF01658872. PMID 2815801
- [Result] Israelsson LA. Parastomal hernias. Surg Clin North Am. 2008 Feb;88(1):113-25, ix. doi: 10.1016/j.suc.2007.10.003. PMID 18267165
- [Result] Martin L, Foster G. Parastomal hernia. Ann R Coll Surg Engl. 1996 Mar;78(2):81-4. PMID 8678463
- [Result] Marimuthu K, Vijayasekar C, Ghosh D, Mathew G. Prevention of parastomal hernia using preperitoneal mesh: a prospective observational study. Colorectal Dis. 2006 Oct;8(8):672-5. doi: 10.1111/j.1463-1318.2006.00996.x. PMID 16970577
- [Result] Etherington RJ, Williams JG, Hayward MW, Hughes LE. Demonstration of para-ileostomy herniation using computed tomography. Clin Radiol. 1990 May;41(5):333-6. doi: 10.1016/s0009-9260(05)81696-4. PMID 2354601
- [Result] Cheung MT, Chia NH, Chiu WY. Surgical treatment of parastomal hernia complicating sigmoid colostomies. Dis Colon Rectum. 2001 Feb;44(2):266-70. doi: 10.1007/BF02234303. PMID 11227945
- [Result] Pastor DM, Pauli EM, Koltun WA, Haluck RS, Shope TR, Poritz LS. Parastomal hernia repair: a single center experience. JSLS. 2009 Apr-Jun;13(2):170-5. PMID 19660211
- [Result] Rubin MS, Schoetz DJ Jr, Matthews JB. Parastomal hernia. Is stoma relocation superior to fascial repair? Arch Surg. 1994 Apr;129(4):413-8; discussion 418-9. doi: 10.1001/archsurg.1994.01420280091011. PMID 8154967
- [Result] Stephenson BM, Phillips RK. Parastomal hernia: local resiting and mesh repair. Br J Surg. 1995 Oct;82(10):1395-6. doi: 10.1002/bjs.1800821033. No abstract available. PMID 7489176
- [Result] Hammond TM, Huang A, Prosser K, Frye JN, Williams NS. Parastomal hernia prevention using a novel collagen implant: a randomised controlled phase 1 study. Hernia. 2008 Oct;12(5):475-81. doi: 10.1007/s10029-008-0383-z. Epub 2008 May 17. PMID 18484151
- [Result] Serra-Aracil X, Bombardo-Junca J, Moreno-Matias J, Darnell A, Mora-Lopez L, Alcantara-Moral M, Ayguavives-Garnica I, Navarro-Soto S. Randomized, controlled, prospective trial of the use of a mesh to prevent parastomal hernia. Ann Surg. 2009 Apr;249(4):583-7. doi: 10.1097/SLA.0b013e31819ec809. PMID 19300232
- [Result] Janes A, Cengiz Y, Israelsson LA. Preventing parastomal hernia with a prosthetic mesh: a 5-year follow-up of a randomized study. World J Surg. 2009 Jan;33(1):118-21; discussion 122-3. doi: 10.1007/s00268-008-9785-4. PMID 19011935
- [Result] Shabbir J, Chaudhary BN, Dawson R. A systematic review on the use of prophylactic mesh during primary stoma formation to prevent parastomal hernia formation. Colorectal Dis. 2012 Aug;14(8):931-6. doi: 10.1111/j.1463-1318.2011.02835.x. PMID 21929523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Ideal Conduit No Mesh | Group 2 - Ileal Conduit With Mesh
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Sponsor Termination | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Ideal Conduit No Mesh | Group 2 - Ileal Conduit With Mesh | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 4 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Rate of Reduction of the Incidence of Parastomal Hernia
Description: Rate of reduction of the incidence of parastomal hernia in study participants, as assessed by physical examination
Time Frame: 18 months
Population: The study required a minimum of 13 participants enrolled per arm for analysis of this outcome measure. Due to the manufacturer's (Ethicon) termination of the Physiomesh device, the study was prematurely terminated with fewer than minimum number of participants required on each arm, and the data were not analyzed.
Arm/Group | Group 1 - Ideal Conduit No Mesh | Group 2 - Ileal Conduit With Mesh
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Who Develop Mesh Related Complications
Description: Assessed by physical examination including:
  * Mesh erosion and infection
  * Stomal stenosis and necrosis
  * Frequency of stoma pouch appliance changes.
  * Record by physical exam the incidence of parastomal hernia at 5 years.
Time Frame: 60 months
Population: as for outcome 1
Arm/Group | Group 2 - Ileal Conduit With Mesh
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1 - Ideal Conduit No Mesh | Group 2 - Ileal Conduit With Mesh
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
This study required a minimum of 13 participants enrolled per arm. Due to the manufacturer's (Ethicon) termination of the Physiomesh device, the study was prematurely closed with fewer than minimum number of participants required per arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes